CLINICAL TRIAL: NCT05215730
Title: Comparison of Wound Healing Efficacy Between MedCu Wound Dressings With Copper Oxide and Negative Pressure Wound Therapy (NPWT/VAC) Treatment
Brief Title: Comparison of Wound Healing Between MedCu Dressings With Copper Oxide and Negative Pressure Wound Therapy Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedCu Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WD-2C-1012-02-IL
Record Dates: First submitted 2022-01-03; First posted 2022-01-31 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Wounds and Injuries; Negative Pressure Therapy; Diabetic Foot Ulcer
Keywords: wound dressings; copper oxide; diabetic ulcers; Negative pressure wound therapy
MeSH Terms: conditions — Wounds and Injuries; Diabetic Foot | interventions — Negative-Pressure Wound Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized multisite two arms study: one arm will be treated with Negative Pressure Wound Therapy (NPWT) known also as Vacuum-assisted closure (VAC) treatment ("VAC Arm"). The second arm with MedCu wound dressings with copper oxide (COD) ("Copper Arm").
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Copper oxide dressings (COD) (Active Comparator): MedCu wound dressings with copper oxide (COD) ("Copper Arm").
  Interventions: Device: MedCu wound dressings with copper oxide (COD)
- Vacuum-assisted closure (VAC) treatment ("VAC Arm") (Active Comparator): Negative Pressure Wound Therapy (NPWT) known also as Vacuum-assisted closure (VAC) treatment ("VAC Arm").
  Interventions: Device: MedCu wound dressings with copper oxide (COD)

INTERVENTIONS:
Device: MedCu wound dressings with copper oxide (COD) — Patients whose foot wound is indicated for VAC treatment will be randomized to either treatment arm after signing informed consent.
  Other Names: Negative Pressure Wound Therapy (NPWT) known also as Vacuum-assisted closure (VAC) treatment

SUMMARY:
Randomized multisite two arms study in which one arm of patients will be treated with Negative Pressure Wound Therapy (NPWT) known also as Vacuum-assisted closure (VAC) treatment ("VAC Arm") and the second arm of patients will be treated with MedCu wound dressings with copper oxide (COD) ("Copper Arm"). The study goals are to compare the efficacy, cost and convenience between MedCu Wound Dressings with Copper Oxide (COD) and Negative Pressure Wound Therapy of diabetic foot wounds.

DETAILED DESCRIPTION:
Randomized multisite two arms study: one arm will be treated with Negative Pressure Wound Therapy (NPWT) known also as Vacuum-assisted closure (VAC) treatment ("VAC Arm"). The second arm with MedCu wound dressings with copper oxide (COD) ("Copper Arm").

Prior to the commencement of the study the patients will be treated according to the caregiver routine and the wound and patient condition, e.g. surgical or bedside debridement, minor foot amputation and/or various wound dressings. Patients whose foot condition has improved and there is indication for VAC treatment will be randomized to either treatment arm after signing informed consent.

The patients will be then treated for 2-8 weeks with the study treatment.

Treatment termination - Treatment will be stopped due to the following reasons:

1. Treatment failure

   1. Wound deterioration
   2. Wound infection
   3. Adverse events
2. Inability to continue the current treatment for any other reason unrelated to the treatment modality
3. Expected termination (two to eight weeks) - no indication to continue treatment arm or if sufficient granulation has been achieved and the patient is candidate for skin grafting
4. Wound closure The VAC treatment will be performed twice weekly, according to the routine practice (usually 75-150 mm Hg). The COD will be changed once a week or more often in highly exudating wounds. The patients will be monitored at least every two weeks in the clinic, but documentation of the wound condition will be obtained in every dressing change or VAC replacement.

Follow-up Period - Patients will be monitored for two additional weekly or biweekly visits (total of 2-4 weeks). The Follow-up Period will be following treatment termination (including wound closure).

In the follow-up period the patient will be treated according to the physician decision based on standard of care, available treatment and wound condition. Continue treatment with the same arm modality, for which the patient had been randomized is allowed and will be recorded. Change into the other arm treatment will be allowed but will be documented as a "Cross Over" and the reason for the cross over will be stated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18 to 85 years of age at the time of enrollment.
2. Subject has Diabetes Mellitus (type 1 or type 2) by WHO criteria.
3. Wounds in which a decision to treat it with Negative Pressure Wound Therapy (NPWT) has been made due to the wound condition and the physician practice (the wound should be one that deem suitable to NPWT treatment).
4. In the case of wounds involving the plantar aspects, they should be without significant bony prominences (unless off-loading can effectively relieve these pressure areas).
5. The wound does not have overt signs of infection or if there is residual infection, it is under control and in the process of resolving as evidenced by laboratory tests (within one day prior to study commencement for in-house patients) and clinical judgment.
6. The wound type configuration and location clearly allows the application of VAC with efficient sealing.
7. If there are additional wounds in the same foot that can be connected by the same VAC apparatus, then each wound will be considered as an index wound and analyzed separately. If there are additional wounds that cannot be connected by the VAC apparatus, the criteria to include the patient in the study is that these wounds can be dressed separately and not interfere with the VAC apparatus. These wounds will be treated by SOC and will not be included in the statistical analysis.
8. Vascular assessment:

   1. All patients need to have ankle-brachia index (ABI) determination even in the presence of palpable pulses. If ABI is > 0.5 in both arteries, or >0.8 in at least one artery, the patient will be eligible to participate in the study.
   2. Patients in whom reliable ABI cannot be obtain due to non-compressible arteries, toe-brachial index (TBI) will be assessed and it needs to be > 40.
   3. Patients who have undergone successful vascular intervention will be assessed by ABI measurements. Nevertheless, if in such patients the value will negate participation in the study, vascular surgeon consultation or interventional radiologist report on good outcome during the procedure will allow inclusion in the study.
9. Having a body mass index (BMI) <45 Kg/m2.
10. Recent glycosylated haemoglobin (HbA1c) <12.0%.
11. Recent creatinine level ≤3.0 mg/dL.
12. No further surgery to handle the wound or the infection is expected or contemplated.
13. The patient is able and eligible to sign written informed consent and participate in the study.
14. Be available for the entire study period, and ability and willingness to adhere to the requirements of the study.

Exclusion Criteria:

1. General conditions:

   * Unstable cardiac disease or other medical conditions with expected repeated hospitalizations during the study phase.
   * Participation in an investigational trial (active phase) at the time of study inclusion.
   * History of allergic reactions attributed to copper; Wilson disease.
   * Any patients receiving or expected to receive chemotherapy during the study period.
   * Any form of substance abuse (including drug or alcohol abuse, excluding cannabis), psychiatric disorder or any chronic condition susceptible, in the opinion of the investigator, of interfering with the conduct of the study.
   * Females who are pregnant, lactating, of child-bearing potential.
   * Fertile female subjects who are not willing to use an acceptable method of contraception during the treatment period and for 14 days following completion of treatment.
   * Subjects who are likely to be non-compliant or uncooperative during the study.
   * Subjects and conditions in which a non-approval of VAC therapy (usually be the HMO) is expected or suspected.
2. Laboratory tests:

   * Anemia (Hemoglobin < 7.0 g/dL).
   * BMI > 45 Kg/m2.
   * White Blood Cells count > 12,000/μL (higher levels are affordable if clinical improvement and other laboratory signs of improvement are evident).
   * Platelet's count < 75,000/μL.
   * Albumin < 2.0 g/dL.
   * CRP - may be higher than normal but should be stable at the time of enrollment or a with a trend toward improvement.
   * Blood Creatinine > 3.0 mg/dL at the time of enrolment.
   * Any other clinically significant blood and urinalysis tests abnormalities that can jeopardize study results as evaluated by the investigator.
3. Wound condition:

   * Any signs of active or residual infection of the wound that need close inspection and/or repeated debridement.
   * Wounds that deem unsuitable to NPWT treatment due to expected problem of sealing the wound (e.g. wound with toe clefts) or too painful to handle such treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Change in wound size | 4, 8 and 12 weeks of treatment
  The size of the wound will be determined by using a 3D Wound Imaging System

SECONDARY OUTCOMES:
Physiological parameter - Change in granulation tissue | 4, 8 and 12 weeks of treatment
  Percentage of granulation tissue will be determined based on the physicians evaluation and by Tissue Analytics Imaging system
Physiological parameter - Percentage of wounds that will be closed during the study period | 12 weeks
  The percent of closed wounds per study group will be calculated and compared
Cost of treatment | 12 weeks
  The mean cost of treatment per patient in each of the two study groups will be calculated. It will include cost of the actual equipment (dressings versus VAC) and time of treatment by caregivers.
Convenience - patient perspective - Questionnaire | 12 weeks
  The patients will be asked to give an indication of their convenience perspective of the treatment by giving a grade between 1-10, being 1 "not convenient at all" and 10 "very convenient".
Convenience - caregiver perspective - Questionnaire | 12 weeks
  The caregivers will be asked to give an indication of their convenience perspective of the treatment by giving a grade between 1-10, being 1 "not convenient at all" and 10 "very convenient".
Pain - patients perspective - Questionnaire | 12 weeks
  The patients will be asked to give an indication of the pain they felt during treatment by giving a grade between 1-10, being 1 "felt no pain" and 10 "felt extreme pain".
Physiological parameter - Infectious episodes | 12 weeks
  The number of infectious episodes, which will include fever, antibiotic administration, and wound infection, during the trial will be recorded and compared between both study arms.
Physiological parameter - Number of treatment-related adverse events as assessed by CTCAE v4.0 | 12 weeks
  The number of treatment-related adverse event episodes during the trial will be assessed in both study arms according to CTCAE v4.0
Physiological parameter - Change in necrotic tissue | 4, 8 and 12 weeks of treatment
  Percentage of necrotic tissue will be determined based on the physicians evaluation and by Tissue Analytics Imaging system
Physiological parameter - Change in fibrin tissue | 4, 8 and 12 weeks of treatment
  Percentage of fibrin tissue will be determined based on the physicians evaluation and by Tissue Analytics Imaging system
Physiological parameter - Average time to wound closure | 12 weeks
  The average time to close the wounds in each arm will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Melamed, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel